CLINICAL TRIAL: NCT03965611
Title: From the Brain to the Bugs: Evolution of Oropharyngeal and Rectal Microbiota of Patients With Severe Traumatic Brain Injury Admitted in ICU
Brief Title: Evolution of Oropharyngeal and Rectal Microbiota After Severe Traumatic Brain Injury
Acronym: BBAX
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Université Paris-Saclay (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180537; 2018-A02973-52 (Other: IDRCB)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury; Multiple Trauma
Keywords: Traumatic brain injury; Multiple trauma; Microbiota; Intensive care unit
MeSH Terms: conditions — Brain Injuries, Traumatic; Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen types :
  * Oropharyngeal swabs
  * Rectal swabs
  The swabs will be performed for each patient within the first 24 hours after ICU admission (day 0), then 48 hours (day 2) and 7 days (day 7) after ICU admission and weekly thereafter until ICU discharge. Rectal and oropharyngeal swabs will be performed by trained paramedical staff using sterile swabs with transport medium ESwab® (Becton, Dickinson and Company, New Jersey, USA). Swabs will be stored at -80°C until bacterial DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with isolated severe traumatic brain injury (TBI): TBI with initial Glasgow Coma Scale (GCS) ≤ 8 and AISextrahead score ≤3. Oropharyngeal and rectal swabs will be performed for each patient within the first 24 hours after ICU admission (day 0), then 48 hours (day 2) and 7 days (day 7) after ICU admission and weekly thereafter until ICU discharge.
  Interventions: Procedure: Oropharyngeal swab; Procedure: Rectal swab; Procedure: Disability rating scale (DRS-F)
- Patients with severe trauma without TBI: Patients with severe trauma without TBI (AISextrahead score > 3). Oropharyngeal and rectal swabs will be performed for each patient within the first 24 hours after ICU admission (day 0), then 48 hours (day 2) and 7 days (day 7) after ICU admission and weekly thereafter until ICU discharge.
  Interventions: Procedure: Oropharyngeal swab; Procedure: Rectal swab; Procedure: Disability rating scale (DRS-F)
- Healthy Controls: Persons who have not had the conditions being studied or otherwise related conditions or symptoms, as specified in the eligibility requirements.
  Oropharyngeal and rectal swabs will be taken only once, at inclusion, after that the participation of the control individual in the trial will be completed.
  Interventions: Procedure: Oropharyngeal swab; Procedure: Rectal swab

INTERVENTIONS:
Procedure: Oropharyngeal swab — Will be performed by trained paramedical staff using sterile swabs with transport medium ESwab® (Becton, Dickinson and Company, New Jersey, USA). Swabs will be stored at -80°C until DNA extraction.
Procedure: Rectal swab — Will be performed by trained paramedical staff using sterile swabs with transport medium ESwab® (Becton, Dickinson and Company, New Jersey, USA). Swabs will be stored at -80°C until DNA extraction.
Procedure: Disability rating scale (DRS-F) — Will be assessed at day 90 +/- 7 days.
  Groups: Patients with isolated severe traumatic brain injury (TBI); Patients with severe trauma without TBI

SUMMARY:
Modifications of the human gut microbiota have been associated with different pathological conditions such as obesity, inflammatory bowel diseases and neurodegenerative diseases. Recently the " Brain-Gut Axis ", a bidirectional communication axis between brain and gut, has been described. In recent animal studies, an acute brain injury was associated with rapid modifications of the gut microbiota.

In humans, traumatic brain injury (TBI) is a leading cause of death and disability. The patterns of gut and oropharyngeal microbiota following TBI are unknown. The primary purpose of this study is to characterize gut and oropharyngeal microbiota of patients with severe TBI.

DETAILED DESCRIPTION:
Study Protocol :

Observational prospective cohort study.

Patients

Patients admitted to the ICU for severe trauma will be included. Two groups of patients with severe trauma will be studied:

1. Patients with isolated severe traumatic brain injury (TBI): TBI with initial Glasgow Coma Scale (GCS) ≤ 8 and AISextrahead score ≤3
2. Patients with severe trauma without TBI (AISextrahead score > 3)

A group of healthy individuals will serve as a control population.

Expected total enrollment 20 patients in each group, and 10 healthy controls.

Patient data collection

For each patient, the following data will be collected:

* Demographic data: age, sex, height, weight, ICU admission date, simplified acute physiology score II (SAPS II), injury severity score (ISS), abbreviated injury scale (AIS) at ICU admission.
* Trauma-related data: number and type of trauma-related organ injuries, initial GCS, presence of mydriasis at initial management.
* Factors with potential impact on microbiota: antimicrobial therapy, nutrition type, medications (proton pump inhibitors, opioids, sedations, catecholamines, steroids), surgical procedure during ICU stay.
* Evolution: multidrug resistant bacteria acquisition during ICU stay, ICU acquired-infections. Mechanical ventilation duration, extrarenal epuration, ICU length of stay, neurological outcome evaluated by disability rating scale (DRS-F) at ICU discharge and at 90 days post trauma, death at ICU discharge and 90 days.

Sample collection

Oropharyngeal and rectal swabs will be performed for each patient within the first 24 hours after ICU admission (day 0), then 48 hours (day 2) and 7 days (day 7) after ICU admission and weekly thereafter until ICU discharge. Rectal and oropharyngeal swabs will be performed by trained paramedical staff using sterile swabs with transport medium ESwab® (Becton, Dickinson and Company, New Jersey, USA). Swabs will be stored at -80°C until DNA extraction.

DNA extraction

DNA extraction will be performed using QIAamp PowerFecal Pro DNA® kit (Qiagen®, Courtaboeuf, France) for rectal swabs and Extracta DNA Prep® kit (Quanta Biosciences®, Beverly, USA) for oropharyngeal swabs. DNA will be quantified by Quantit® dsDNA HighSensitivity Assay Kit (Fisher Scientific).

16S rRNA amplification and sequencing

V3 and V4 regions of bacterial 16S rRNA gene sequences will be amplified by polymerase chain reaction (PCR) with universal primers (TCGTCGGCAGCGTCAGATGTGTATAAGAGACAGCCTACGGGNGGCWGCAG and GTCTCGTGGGCTCGGAGATGTGTATAAGAGACAGGACTACHVGGGTATCTAATCC), following the Illumina MiSeq® System protocol (Illumina®). Amplicons will be purified and then sequenced using MiSeq® sequencing system ((Illumina®).

Sequences processing

Sequences processing and operational taxonomic unit (OTU) clustering will be performed using SHAMAN software (SHiny Application for Metagenomic ANalysis) based on R® software (package DESeq2), provided by Pasteur Institute. Taxonomic classification will be performed using SILVA database reference.

Statistical analysis

Statistical analysis will be performed using SHAMAN software (SHiny Application for Metagenomic ANalysis). Bacterial phyla, families and genera repartition will be analyzed, and relative abundance of bacterial genera will be compared between the different populations. Alpha-diversity will be analyzed using different parameters (Shannon index, Simpson's diversity index), as well as beta-diversity (principal component analysis).

The different populations of patients and healthy volunteers will be compared, and the evolution of microbiota along time will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Bicêtre Hospital Trauma Center for severe trauma with:

either isolated severe traumatic brain injury (TBI): TBI with initial Glasgow Coma Scale (GCS) ≤ 8 and AISextrahead score ≤3; either severe trauma without TBI (AISextrahead score > 3)

* Estimated ICU length of stay 48 hours or more

Exclusion Criteria:

* Antimicrobial therapy within the previous 3 months
* Long-term corticosteroids use
* Active cancer
* Institutionalized patient
* Gastro-intestinal perforation or emergency gastro-intestinal surgery following trauma
* Withdrawal of consent
* Patient under guardianship
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years of age or older, admitted to intensive care unit for severe trauma.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in microbiota alpha-diversity as measured by Shannon index | From day 0 to day 90
  The oropharyngeal and rectal swabs, performed at day 0, day 2, day 7 after ICU admission and weekly thereafter until ICU discharge or no later than day 90, will be used for DNA extraction and the bacterial 16S rRNA amplification and sequencing in order to identify the bacterial species colonizing the gut.

SECONDARY OUTCOMES:
Alpha and beta-diversities of oropharyngeal and rectal microbiota at different times post trauma. | From day 0 to day 90
  The oropharyngeal and rectal swabs, performed at day 0, day 2, day 7 after ICU admission and weekly thereafter until ICU discharge or no later than day 90, will be used for DNA extraction and the bacterial 16S rRNA amplification and sequencing in order to identify the bacterial species.
ICU-acquired infections | From day 0 to day 90
  The ICU-acquired infection rates during the ICU stay
Number of patients acquiring colonization or infection with multidrug resistant bacteria during ICU stay | From day 0 to day 90
  Multidrug resistant bacteria colonisation or infection acquired during the ICU stay
Death at ICU discharge and 90 days post trauma. | From day 0 to day 90
  The rates of deaths at ICU discharge and 90 days post trauma
Disability Rating Scale (DRS-F) score at 90 days post trauma | From day 0 to day 90
  Neurological outcome at 90 days post trauma evaluated by the Disability Rating Scale, the French translation (DRS-F) quoted from 0 (no disability) to 29 (extreme vegetative state)

CONTACTS AND LOCATIONS:
Overall Officials: Samy Figueiredo, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- APHP Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided